CLINICAL TRIAL: NCT02943486
Title: Mesenchymal Stromal Cell Derivatives: a New Alternative and Potential Product for the Treatment of Diabetic Foot Ulcers 1 and 2
Brief Title: Mesenchymal Stromal Cell Derivatives in the Treatment of Chronic Diabetic Foot Ulcers Type 1 and 2
Acronym: MSCDTDFU
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad Autónoma de Bucaramanga (Other)
Collaborators: Fundación Oftalmológica de Santander Clínica Carlos Ardila Lulle (Other); Instituto Colombiano para el Desarrollo de la Ciencia y la Tecnología (COLCIENCIAS) (Other Government)
Responsible Party: Principal Investigator, Claudia Lucia Sossa Melo, Associate Professor, Universidad Autónoma de Bucaramanga
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 124174455522
Record Dates: First submitted 2016-10-19; First posted 2016-10-24 (Estimated); Last update posted 2016-10-24 (Estimated); Status verified 2016-10

CONDITIONS: Foot Ulcer, Diabetic
Keywords: Mesenchymal stromal cells; Fitostimoline; MSC derivatives; Diabetes
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus | interventions — Cell- and Tissue-Based Therapy; Flour

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- dac-MSCs and Fitostimoline (Experimental): Intradermic application of dac-MSCs (1 mL ) in four equidistant points around the ulcer (twice: day 0 and 7) and topical application of fitostimoline every other day
  Interventions: Other: dac-MSCs; Drug: Fitostimoline
- MSCs and Fitostimoline (Active Comparator): Intradermic application of MSCs (500,000 cells/mL) in four equidistant points around the ulcer (once: day 0 ) and topical application of fitostimoline every other day
  Interventions: Other: MSCs; Drug: Fitostimoline
- Fitostimoline (Active Comparator): Topical application of fitostimoline every other day
  Interventions: Drug: Fitostimoline

INTERVENTIONS:
Other: dac-MSCs — Cell-free therapy
  Other Names: Cell-free therapy
  Arms: dac-MSCs and Fitostimoline
Other: MSCs — Cell-based therapy
  Other Names: Cell-based therapy
  Arms: MSCs and Fitostimoline
Drug: Fitostimoline — Triticum vulgare
  Other Names: Triticum vulgare

SUMMARY:
The goal of this study is to evaluate the safety and efficacy of using mesenchymal stromal cell derivatives (dac-MSCs) in the treatment of chronic diabetic foot ulcers (type 1 and 2) in adults. A third of the participants will receive dac-MSCs and Triticum vulgare (Fitostimoline) in combination, the other third MSCs and Fitostimoline in combination, and the last third only Fitosimoline. This study will be a randomized, blind, and parallel and controlled-group trial.

DETAILED DESCRIPTION:
Conventional treatments such as dry, wet or active dressings are effective only in 50% of patients with diabetic foot ulcer. The remaining 50% of patients have non-responding recoveries that leads to amputation of the compromised limbs. Currently, the administration of mesenchymal stem cells (MSCs) in animal models or in small groups of patients with diabetic foot ulcer has shown to be safe and effective. Particularly, the use of these cells induce regeneration, both in the dermis and the epidermis. Nevertheless, MSC transplantation has some limitations, for instance, time restrictions in the availability of cells due to their isolation and expansion as well as the complex and costly large-scale production. In the same manner, the cryopreservation might cause deleterious effects that affect the biological activity of the cells and a medical professional should conduct the cell administration. In addition, different studies report variability in the results due to the inconsistency in the methods that they used (extraction protocols, cultivation, expansion and administration). The investigators' recent studies in mice with skin lesions, particularly type 1 diabetes, have shown that the presence of the cells is not necessary to promote skin regeneration and the administration of dac-MSCs is sufficient to stimulate would healing.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between the ages of 40 and 80 years, inclusive, with Type 1 or 2 diabetes as defined by the American Diabetes Association
* Stable glycemic control
* Transcutaneous oxygen measurement > 30 mmHg
* Ulcer present at least for 1 month
* Wound size between 0.5 and 5 cm2
* Subjects that require endovascular surgical intervention
* Subjects must have adequate nutrition (albumin level > 2 g/dL and prealbumin level > 15 mg/dL)

Exclusion Criteria:

* Previous or current diagnoses with one of the following: cancer, symptomatic coronary artery disease, brain disease, kidney failure, blood disorders
* Taking immunosuppressive and cytotoxic drugs
* Presence of active systemic infection

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2017-01; Primary Completion 2018-06 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Wound size change | One year
  Wound size will be assessed using a SilhouetteMobile camera (digital planimetry)

SECONDARY OUTCOMES:
Granulation tissue percentage | One year
  Images will be used to assess the amount of granulation tissue present in the wound
Pigmentation change | One year
  Digital images will be used to evaluate color changes in the wound
Presence of Exudate | One year
  Visual observation of the wound to determine the presence of exudate

CONTACTS AND LOCATIONS:
Overall Officials: Claudia L Sossa-Melo, MD, Principal Investigator — Universidad Autónoma de Bucaramanga

IPD SHARING:
Plan to Share IPD: No